CLINICAL TRIAL: NCT05526001
Title: A Phase III, Randomized, Parallel, Double-blinding, 2-Arm Study to Investigate the Efficacy and Safety of Intra-articular ELIXCYTE (Adipose-Derived Stem Cells) Injection Compared With Placebo in Subjects With Knee Osteoarthritis
Brief Title: Efficacy and Safety of ELIXCYTE Intra-articular Injection in Subject With Knee Osteoarthritis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UnicoCell Biomed CO. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT22
Record Dates: First submitted 2022-08-28; First posted 2022-09-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ELIXCYTE (Experimental): Subjects will be intra-articular (IA) injected with 4 mL of ELIXCYTE (containing 32×10^6 ADSCs) at the target knee once
  Interventions: Biological: ELIXCYTE
- Placebo control (Saline) (Placebo Comparator): Subjects will be intra-articular (IA) injected with 4 mL of saline at the target knee once
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: ELIXCYTE — ELIXCYTE, a new investigational product developed by UnicoCell Biomed, contains allogenic Adipose-derived stem cells (ADSCs). The ADSCs of ELIXCYTE for subjects were obtained from donors, and the Sponsor followed the manufacturing and testing procedures described in chemistry, manufacturing and control (CMC) information in order to assure the quality of final products.
  Arms: ELIXCYTE
Drug: Saline — Placebo control used in the study.
  Arms: Placebo control (Saline)

SUMMARY:
This is a Phase III, double-blinded, placebo-controlled, multicenter study to investigate the efficacy and safety of a new study intervention, ELIXCYTE, compared to placebo (normal saline) in subjects with knee osteoarthritis. The primary hypothesis of the study is to demonstrate that ELIXCYTE is superior to placebo (saline) in improving knee pain on the target knee from baseline.

During the study, each participant will receive either ELIXCYTE (study intervention) or placebo (normal saline) intra-articular injection once on the target knee after eligibility criteria check. The target knee will be assessed by X-ray, MRI and subject self-evaluation knee questionnaires (WOMAC, KSS and KOOS) in the following visits. Other safety assessments, including lab test, physical examination, vital sign, medical/medication history and adverse events will also be collected throughout the study.

DETAILED DESCRIPTION:
This Phase III study is a prospective, double-blind, parallel, multicenter, 2-arm study to evaluate the efficacy and safety of intra-articular ELIXCYTE injection compared to placebo in subjects with knee OA. All the subjects will be enrolled in Taiwan. Subjects aged 40 to 80 years with knee OA will be enrolled in the study. Approximately 165 eligible subjects will be randomized to receive either ELIXCYTE, or placebo in a 2:1 ratio.

The target population will be composed of subjects with unilateral or bilateral knee OA. For subjects with bilateral OA knees, only the knee with more severe symptoms will be selected as the target knee, while the non-target knee can continue the regular local treatment for ethical consideration. If the severities of the OA symptoms will be the same for both knees, the knee with more pain should be selected based on the WOMAC pain score. Eligible subjects will be randomized into one of the study groups (ELIXCYTE, or placebo in a 2:1 ratio).

The study consists of 9 visits and the duration per subject will be approximately 50 weeks (14 days of screening period, a treatment visit on Day 1, and 48 weeks of evaluation period). Unscheduled visit(s) may be arranged when deem necessary by the investigator.

In addition, if ELIXCYTE provided medical benefits with no safety issues to ELIXCYTE group at the end of week 48, subjects assigned to placebo group will be offered a treatment with ELIXCYTE under an extension study after study unblinding.

ELIGIBILITY:
Inclusion Criteria:

A subject is eligible for the study if all of the following apply:

1. Either gender, aged 40 to 80
2. With unilateral/bilateral knee OA of Kellgren-Lawrence grading II-III (determined by American College of Rheumatology criteria of knee OA).
3. WOMAC pain score of 7 - 17 in the target knee even if treated with chronic doses of NSAID.
4. Has received 1 - 3 types of pharmacological therapies for knee OA for more than 3 months but the symptoms have not relieved.
5. Unwilling or not suitable to undergo knee surgery (including total knee replacement and knee arthroplasty).
6. Understands and has signed the informed consent form.
7. With adequate hematological indices:

   * White blood cell (WBC) ≥ 3,000/mm3
   * Platelet count ≥ 80,000/μL
8. With adequate coagulation indices: Prothrombin time (PT), international normalized ratio (INR), and activated partial thromboplastin time (APTT) ≤ 1.5 times the upper limit of the normal range (ULN).
9. With adequate liver function where serum total bilirubin ≤ 1.5 times ULN, aspartate aminotransferase (AST) ≤ 3 times ULN, and alanine aminotransferase (ALT) ≤ 3 times ULN.
10. Has an estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73m2, calculated by the Modification of Diet in Renal Disease (MDRD) equation.

Exclusion Criteria:

Any subject meeting any of the exclusion criteria will be excluded from study participation.

1. With previous surgery of articular fracture, ligament reconstruction, meniscal reconstruction (with the exception of meniscal debridement), and knee arthroplasty on the target knee joint.
2. With any IA intervention of the target knee within 3 months prior to screening (e.g. steroid, anesthetic), or sodium hyaluronate by IA intervention of the target knee within 6 months prior to screening.
3. Administered systemic immunosuppressive agent, systemic antiinflammatory drug, systemic steroid, systemic analgesics (except acetaminophen, and tramadol as rescue medications), duloxetine, or over-the-counter medications contain analgesics (e.g. cold medicine) within 2 weeks prior to screening. Administered systemic herbal, homeopathic, or naturopathic remedies for knee OA within 2 weeks prior to screening. A subject requiring routine use of low-dose Aspirin for preventing thrombosis (≤ 100 mg/day) will not be excluded from this study
4. Administered local immunosuppressive agent, local anti-inflammatory drug, local steroid, local analgesics, over-the-counter medications contain analgesics, herbal, homeopathic, or naturopathic remedies for knee OA within 2 weeks prior to screening.
5. Has participated in other investigational studies within 4 weeks prior to screening.
6. Administered monoamine oxidase inhibitor, selective serotonin reuptake inhibitor, serotonin-norepinephrine reuptake inhibitors, benzodiazepine, or tricyclic antidepressants within 4 weeks prior to screening.
7. With joint diseases expect knee OA that is considered not eligible to enter the study by the investigator.
8. Systemic diseases that may affect joints, including but not limited to inflammatory joint diseases, reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, and fibromyalgia.
9. Known or suspected infection around the target knee joint.
10. Has serious medical conditions or ongoing disease (e.g. concomitant illness such as cardiovascular (e.g. New York Heart Association grade III or IV), hepatic (e.g. Child-Pugh Class C), psychiatric condition, alcoholism, drug abuse), medical history, physical findings, or laboratory abnormality that in the investigators' opinion could interfere with the results of the trial or adversely affect the safety of the subject.
11. With any evidence of malignant disease with a life expectancy less than 1 year.
12. With a known history of human immunodeficiency virus (HIV) infection.
13. With a known history of alcohol abuse.
14. With a known history of opioid dependent.
15. Known or suspected hypersensitivity to any ingredients of the investigational product (ELIXCYTE) or contrast medium for magnetic resonance imaging (MRI).
16. Body mass index (BMI) ≥ 35 kg/m2
17. Judged to be not applicable to this study by investigator such as the difficulty of follow-up observation.
18. Has claustrophobia and/or cannot take MRI test.
19. Has any existing active/inactive implanted medical devices that pose a safety risk during MRI examination, such as a cardiac pacemaker, cochlear, intracranial vascular clips, or neurostimulator, etc.
20. Has any existing metallic intraocular foreign body that pose a safety risk during MRI examination.
21. Female subject of childbearing potential who:

    * Is lactating; or
    * Has positive pregnancy test result at eligibility checking; or
    * Refuses to adopt at least one form of birth control from signing informed consent to the end of the study.
22. Male subject with female spouse/partner who is of childbearing potential refuses to adopt at least one form of birth control from signing informed consent to the end of the study.
23. Known allergy to acetaminophen and tramadol.
24. Has any abnormal radiographic evidence of target knee, such as excessive malalignment, other arthropathies, or systemic metabolic bone disease, etc.
25. Known any contraindication to IA intervention of the target knee, such as skin infection of injection site, coagulopathy, or routine use of anticoagulant, etc.

For exclusion criteria #21 and #22, acceptable forms of birth control include:

* Established use of oral, injected, or implanted hormonal methods of contraception.
* Placement of an intrauterine device (IUD) or intrauterine system (IUS).
* Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change of WOMAC pain score on the target knee | Baseline, Week 24
  WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) is a questionnaire to evaluate the condition of subjects with knee OA. The pain score ranges from 0 to 20.

SECONDARY OUTCOMES:
Percentage of pain responders (WOMAC pain score) | Week 24 and Week 48
  The responders are defined as subjects who had at least a 20% reduction in WOMAC pain score from baseline.
Total scores of WOMAC | Screening visit, Day 1, Week 2, 4, 12, 24, 36 and 48
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a standardized questionnaire to evaluate the condition of subjects with knee OA in terms of pain, stiffness, and physical functioning of the joints. It contains 5 items for pain (score range 0 ~ 20), 2 for stiffness (score range 0 ~ 8), and 17 for functional limitation (score range 0 ~ 68). The total score of the question ranges from 0 to 96
Pain subscale of WOMAC | Screening visit, Day 1, Week 2, 4, 12, 24, 36 and 48
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a standardized questionnaire to evaluate the condition of subjects with knee OA in terms of pain, stiffness, and physical functioning of the joints. It contains 5 items for pain, and the total pain score ranges from 0 to 20.
Stiffness subscale of WOMAC | Screening visit, Day 1, Week 2, 4, 12, 24, 36 and 48
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a standardized questionnaire to evaluate the condition of subjects with knee OA in terms of pain, stiffness, and physical functioning of the joints. It contains 2 items for stiffness, and the total stiffness score ranges from 0 to 8.
Functional subscale of WOMAC | Screening visit, Day 1, Week 2, 4, 12, 24, 36 and 48
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a standardized questionnaires to evaluate the condition of subjects with knee OA in terms of pain, stiffness, and physical functioning of the joints. It contains 17 items for functional limitation, and the total functional score is ranging from 0 to 68.
Visual Analogue Scale (VAS) for pain | Screening visit, Day 1, Week 2, 4, 12, 24, 36 and 48
  Visual analog scale (VAS) is a scale of 100 mm in length to measure subject's pain intensity.
Objective knee score of Knee Society Knee Scoring System (KSS) | Screening visit, Day 1, Week 2, 4, 12, 24, 36 and 48
  The Knee Society Knee Scoring System (KSS) is a system that combines both objective physician-derived and subjective patient-derived component to evaluates OA knee. Five components are included: (1) patient demographics, (2) objective knee score, (3) patient expectation, (4) patient satisfaction, and (5) functional knee score. The objective knee score of KSS includes surgeon part with maximum 75 points and patient self-evaluation part with maximum 25 points.
Functional knee score of Knee Society Knee Scoring System (KSS) | Screening visit, Day 1, Week 2, 4, 12, 24, 36 and 48
  The Knee Society Knee Scoring System (KSS) is a system that combines both objective physician-derived and subjective patient-derived component to evaluates OA knee. Five components are included: (1) patient demographics, (2) objective knee score, (3) patient expectation, (4) patient satisfaction, and (5) functional knee score. The total score of functional knee score ranging from 0 to 100.
Total score of Knee Injury and Osteoarthritis Outcome Score (KOOS) | Screening visit, Day 1, Week 2, 4, 12, 24, 36 and 48
  Knee injury and osteoarthritis outcome score (KOOS) is a questionnaire to assess the patient's opinion about their knee and associated problems. It contains 42 questions and each question is assigned with five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems). The total score of the question ranging from 0 to 168.
Total score of Whole-Organ Magnetic Resonance Imaging Score (WORMS) | Screening, Week 24 and Week 48
  The Whole-Organ-MRI Scores (WORMS) evaluates articular cartilage lesions in 14 anatomic compartments from magnetic resonance imaging (MRI) of the knee by an independent radiologist. Each compartment is scored by 8-point scale (0, 1, 2, 2,5, 3, 4, 5 and 6) and the total score is ranging from 0 to 84.
Cartilage thickness in the total femorotibial joint | Screening, Week 24 and Week 48
  The cartilage thickness will be evaluated by knee MRI
Percentage of subjects using the rescue medication(s) | Screening, through Day 1 to Week 24, through Day 1 to Week 48
  Rescue medication(s) is defined as acetaminophen, and/or tramadol used during the study.
Total used amount of rescue medications used | Screening, through Day 1 to Week 24, through Day 1 to Week 48
  Rescue medication(s) is defined as acetaminophen, and/or tramadol used during the study.
Number of days of rescue medications consumption | Screening, through Day 1 to Week 24, through Day 1 to Week 48
  Rescue medication(s) is defined as acetaminophen, and/or tramadol used during the study.
Time to the first consumption of rescue medications after treatment | through study completion, an average of 1 year
  Rescue medication(s) is defined as acetaminophen, and/or tramadol used during the study.
Incidence of Adverse event (AE) and serious adverse event (SAE) | through study completion, an average of 1 year
  AE means any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product or intervention and which does not necessarily have a causal relationship with this treatment. A SAE is an AE in the view of either the investigator or Sponsor results in any of the following outcomes: death, life-threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect or the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above by medical judgement.
Incidence of AE of special interest (AESI) | through study completion, an average of 1 year
  AEs of special interest (AESI) includes arthralgia, injection site joint pain, injection site joint swelling, and joint swelling.
Incidence of immediate AE | Day 1
  Any adverse event that happens within 30 minutes post-administration of ELIXCYTE or placebo will be considered as an immediate adverse event.
Number of subjects with abnormal vital signs | Screening Visit, Day 1, Week 2, 4, 12, 24, 36 and 48
  Vital signs measurement will consist of respiratory rate, pulse rate, systolic/diastolic blood pressure, and body temperature.
Number of subjects with abnormal findings in laboratory tests | Screening Visit, Day 1, Week 2, 4, 12, 24, 36 and 48
  The laboratory examination includes hematology, biochemistry, immunogenicity and pregnancy tests.
Number of subjects with abnormal findings in physical examination | Screening Visit, Day 1, Week 2, 4, 12, 24, 36 and 48
  The physical examination items include general appearance, skin, eyes, ears, nose, throat, head and neck, heart, chest and lungs, abdomen, extremities, lymph nodes, musculoskeletal, neurological, other body systems if applicable for describing the status of the subject's health.

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Taipei Medical University Shuang-Ho Hospital, New Taipei City, Taiwan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided